CLINICAL TRIAL: NCT07065929
Title: Impact of Early, Personalized Nutritional Management on 1-month Mortality After Acute Stroke Pragmatic, Controlled, Multicenter, Cluster-randomized Trial
Brief Title: Impact of Early, Personalized Nutritional Management on 1-month Mortality After Acute Stroke
Acronym: AVC-NUT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC23_0302; 2025-A00234-45 (Other: ANSM)
Record Dates: First submitted 2025-05-27; First posted 2025-07-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke
Keywords: acute stroke; early nutrition; personalized dietary support
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: cluster randomisation in parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): early nutritional management
  Interventions: Dietary Supplement: Early nutritional management
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Early nutritional management — The food ingested by patients is collected until the day 7 of the stroke so that dieticians can calculate their needs and provide a suitable diet. If this is not sufficient, a reinforced nutrition strategy (meal enrichment) is implemented.
  On day 5 of the stroke, if energy intake is less than 2/3 of the energy objectives, the strategy is switched to level 2, unless it is possible to increase intake within 48 hours.
  Arms: Interventional Group

SUMMARY:
This study evaluate the impact of early personalized nutritional management on 1-month mortality after acute stroke.

In the randomised centres of the interventional group (early personalized nutritional management), each patient will be assessed by a dietician within 2 days of stroke. Any swallowing problems are screened, and any barriers to eating are identified before dietary support. Patient's food intakes are recorded until the 7th day post-acute to assess their energy intake. Depending on patient's nutritional objectives, a reinforced feeding strategy comprising 2 levels is put in place, in order to prevent malnutrition: in level 1, the dietician tries to meet nutritional requirements orally, while in level 2 he can recourse to artificial nutrition in the event of failure or inability to meet requirements with oral intake alone. This strategy is started immediately after the initial assessment. Intakes are reassessed every 24 to 48 hours by the dietician in order to adapt the nutritional strategy as quickly as possible in order to cover the patient's personnalized nutritional needs.

No change in practice was required of the randomised centres in the control group.

All patients will be contacted by telephone 30 days after stroke to collect parts of the assessment criteria, while the other criteria will be collected directly from the patient's computerised medical record.

Three months after stroke, an evaluation of quality of life and modified Rankin test will be performed.

Our hypothesis is that the implementation of an individualized management of early nutritional support, aimed at compensating for the decrease in intake associated with the disease, would reduce mortality at 30 days in patients hospitalised for stroke.

ELIGIBILITY:
Inclusion Criteria :

* Patients ≥ 18 years of age
* With an acute, ischaemic or haemorrhagic outpatient or inpatient stroke
* NIHSS score ≥ 5
* Hospitalised in a neurology department, or Neuro Vascular Unit (NVU), or in a department where beds are dedicated to receiving post-stroke patients
* Stroke less than 2 days old
* Anticipated length of hospital stay in a participating centre ≥ 5 days
* Patient affiliated to or benefiting from a social security scheme
* Patient or close relative having given written consent to participate in the study or patient included under the emergency procedure in the absence of contactable relatives

Exclusion Criteria:

* Patients treated with nutritional therapy at the time of admission (history of bariatric surgery or gastrectomy, malabsorptive pathologies such as short bowel, extensive intestinal resections, etc.).
* In a palliative situation where life expectancy is < 3 months
* Patient taking part in another study with an impact on mortality or nutrition
* Previous inclusion in the trial
* Pregnant, breast-feeding or parturient woman
* Patient unable to follow the protocol for any reason
* Patient deprived of liberty by judicial or administrative decision
* Patient under compulsory psychiatric care
* Person under legal protection
* Poor understanding of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3084 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
mortality at 30 days after stroke (main criterion) | At 30 days of the day of the stroke
  Recording patient status at 30 days after stroke

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin score ≤ 2, 3 months after stroke | At 90 days of the day of the stroke
  Modified Rankin score is evaluated at 3 months after stroke and a percentage of patients with a score < 2 will be calculated
Nutritional status at 30 days defined by BMI, weight change over 30 days and albumin rate, used to classify patients as severely undernourished, moderately undernourished or not undernourished. | At 30 days of the day of the stroke
Time to occurrence of inhalation pneumonia related to the presence of a feeding tube recorded within 30 days of the day of the stroke | Within 30 days of the day of the stroke
  Recording of inhalation pneumonia related to the presence of a feeding tube
Time to occurrence of infection related to a catheter dedicated to parenteral nutrition recorded within 30 days of the day of the stroke | Within 30 days of the day of the stroke
  Recording of infection related to a catheter dedicated to parenteral nutrition
Time to occurrence of death recorded within 30 days of the day of the stroke: | Within 30 days of the day of the stroke
  Recording of death
Hospital stay (in days) with censoring at 3 months after stroke | Length of hospitalization (in days), calculated between the stroke 's date (day 0) and the date of discharge from the Neurology Department, assessed up to 90 days after the stroke.
  Calculation of the number of days of hospitalisation between the stoke and the date of discharge from the Department
Evaluation of the variation in the EuroQol 5D quality of life score (EQ-5D-5L) between the pre-stroke period and 3 months after stroke | At 90 days of the day of the stroke
  Estimated quality of life scores before the stroke and at 3 months post-stroke are obtained using EuroQol 5D-5L questionnaires completed with patients or their close relative at 3 month after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Angélique CAMPION, Principal Investigator — University Hospital, Angers
Locations (12):
- France (12):
  - CH Versailles, Chesnay, Yvelines
  - CHU Angers, Angers
  - CHU Caen, Caen
  - CH Cholet, Cholet
  - CHD La Roche sur Yon, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH Chartres, Le Coudray
  - CHU Rouen, Rouen
  - CHU Nantes, Saint-Herblain
  - CH St Malo, St-Malo
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).